CLINICAL TRIAL: NCT06546319
Title: Music Therapy to Address Patients' Journeys With Chronic Illness, Outcomes, and Readmission (MAJOR CHORD RCT): A Randomized Controlled Trial
Brief Title: Music Therapy to Address Patients' Journeys With Chronic Illness, Outcomes, and Readmission - MAJOR CHORD RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Rodgers-Melnick (Other)
Collaborators: Kulas Foundation (Other)
Responsible Party: Sponsor-Investigator, Samuel Rodgers-Melnick, MPH, MT-BC, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20240686
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Music Therapy; Chronic Obstructive Pulmonary Disease; Heart Failure; In-person; Virtual
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: This study will utilize a mixed-methods intervention design in which qualitative data are embedded in the framework of a randomized controlled trial. Participants receiving music therapy will be compared to participants in a waitlist control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Therapy (Experimental): Participants will complete a series of questionnaires after enrolling, 15 days post hospital discharge, and 30 days post hospital discharge. Board-certified music therapists (i.e., MT-BC credential) will provide two music therapy sessions, not to occur on the same day, that include education and disease-specific content (e.g., harmonica exercises for respiratory health [COPD] or music-based breathing exercises [HF]) prior to patients' discharge and two virtual music therapy sessions that address music-assisted relaxation and imagery, additional techniques for managing psychosocial stressors, and gratitude exercises post-discharge.
  Interventions: Behavioral: Music Therapy
- Control (No Intervention): No additional intervention will be conducted for this arm during their study participation. Participants will complete a series of questionnaires after enrolling, 15 days post hospital discharge, and 30 days post hospital discharge. Participants randomized to the control arm will be offered a single virtual music therapy session after 30 days post-discharge. No data will be collected during this music therapy session.

INTERVENTIONS:
Behavioral: Music Therapy — Board-certified music therapists (i.e., MT-BC credential) will provide two music therapy sessions, not to occur on the same day, that include education and disease-specific content (e.g., harmonica exercises for respiratory health [COPD] or music-based breathing exercises [HF]) prior to patients' discharge and two virtual music therapy sessions that address music-assisted relaxation and imagery, additional techniques for managing psychosocial stressors, and gratitude exercises post-discharge.
  Arms: Music Therapy

SUMMARY:
Conduct a randomized trial (n = 60: with n = 30 receiving music therapy and n = 30 receiving usual care) to investigate the feasibility, acceptability, and preliminary efficacy of the MAJOR CHORD music therapy intervention compared to usual care on (a) health-related quality of life (e.g., physical function, depression, anxiety, fatigue, and pain interference), (b) perceived stress, (c) self-efficacy, and (d) 30-day readmission rates

DETAILED DESCRIPTION:
For the intervention arm, in-person sessions will be conducted at the discretion of the music therapist and at a convenient time for the participant. Post-discharge music therapy sessions will be conducted virtually via secure telehealth platform (i.e., Zoom for Healthcare) with participants at home, skilled nursing facility, or in the hospital, if readmitted, while the music therapist is stationed at UHCMC or another UH facility in a private location. Reminder phone calls and MyCap messages will be completed one day prior to the scheduled virtual session. Links to the virtual session will be sent at the time of scheduling and again just prior to the session.

For both arms, follow-up measures will be completed using REDCap surveys sent via Twilio text message at 15- and 30-days following the hospital discharge date. REDCap will be used to collect the PROMIS - 29, Perceived Stress Scale - 4 (PSS-4), PROMIS General Self-Efficacy 4a, PROMIS Instrumental Support 4a, and PROMIS Emotional Support 4a scores at (1) Baseline, (2) 15-days post discharge, and (3) 30-days post discharge, with REDCap ensuring these are delivered on the nearest weekday rather than a weekend. Reminder texts will be sent out at day 16 & 17 and day 31 & 32 for those who do not complete their follow-up assessments following the initial prompt.

Board-certified music therapists (i.e., MT-BC credential) will provide two music therapy sessions, not to occur on the same day, that include education and disease-specific content (e.g., harmonica exercises for respiratory health [COPD] or music-based breathing exercises [HF]) prior to patients' discharge and two virtual music therapy sessions that address music-assisted relaxation and imagery, additional techniques for managing psychosocial stressors, and gratitude exercises post-discharge. Each music therapy session will include (1) setting an agenda; (2) an explanation of the music exercise; (3) a demonstration of the music exercise in which the MT-BC will engage the participant in practicing the music exercise (e.g., breathing, imagery, harmonica exercise); (4) time to process the participant's response to the exercise; (5) time for the MT-BC to electronically deliver the music exercise to the participant and ensure that the participant has all materials necessary to use the exercise at home; and (6) a homework assignment for the participant to practice the music exercise taught in that session at least once per day until the following MT session. The genres of each music exercise will be personalized to participants' preferences (e.g., hip-hop, gospel, R&B, jazz, rock, and/or soul). Each music exercise will last an average of 12 minutes. As the music exercises are being demonstrated, the MT-BC will simultaneously record the exercise as it is being delivered live. These recordings will be created in a high-quality recording studio, using either (1) a mobile unit in the participant's hospital room during in-person sessions or (2) a virtual music therapy studio at UH Cleveland Medical Center or the music therapist's private office at another UH facility during virtual sessions while participants are at home or in a care facility. The participant will hear the music live and receive a recording at the end of each session for their homework assignment. Each participant's voice may be recorded as part of the second virtual music therapy intervention (i.e., fourth of four sessions) which features a personalized songwriting intervention to which the patient can choose to contribute their voice. These recordings will be uploaded to a personalized UH Enterprise Box folder created for each participant. In-person MT sessions will be audio-recorded, and virtual sessions will be audio and video recorded through UH Zoom for Healthcare for quality assurance and fidelity checking. Recordings will be uploaded to a password-protected secure server and removed from recording devices. MT sessions will be reviewed for quality assurance for the first 5 participants and every 5th participant thereafter.

At the request of the participant, study staff may meet with the participant either in-person prior to discharge or virtually post-discharge to assist the participant in accessing Zoom and practicing the skills needed for videoconferencing (e.g., joining audio, muting, unmuting).

Participants will receive text message links every 7 days following the first music therapy session to log their home exercise activity.

The study staff will coordinate with the participant, participant's family and/or home care nursing team to facilitate the participant's engagement in virtual visits following discharge and before the first virtual music therapy session. The music therapist will provide instructions for virtual access and resources. The study staff will follow up with the participant following discharge to assist them with engaging in virtual music therapy post-discharge.

ELIGIBILITY:
Randomized Control Trial

Inclusion Criteria:

1. Age range: ≥30 to ≤89 years
2. Primary indication for current hospitalization is either COPD or HF with confirmed ICD-10 code in the electronic health record (EHR)
3. Able to read and understand English
4. Hospitalized at UH Cleveland Medical Center (UHCMC) with anticipated length of stay following recruitment ≥ 2 days as documented in electronic health record (EHR) and confirmed by the clinical care team
5. Access to Wi-Fi, active email address, & laptop, tablet, smartphone, and/or PC with videoconferencing capabilities at home or the facility in which they will be discharged
6. Has reliable access to a mobile device with an active data plan at the hospital and at home and is comfortable accessing the internet and their email with this device

Qualitative Interview Inclusion Criteria 1. Agreed to be contacted for the qualitative interview during contenting process for the RCT

Exclusion Criteria:

1. Active confirmed or suspected COVID-19, or under droplet, contact, MRSA, and/or C.diff precaution notification as documented in the EHR
2. Included on the Music Therapy Referral patient list in the EHR
3. Significant hearing and/or visual impairment as documented in EHR
4. Unable to independently provide consent (i.e., no proxy consent)
5. Active suicidal ideation as documented in EHR during current hospital admission
6. Severe psychological comorbidity (e.g., psychosis, schizophrenia) that would prevent patient from engaging fully in intervention as documented in EHR
7. Receiving active cancer treatment (e.g., chemotherapy, radiation, immunotherapy) as documented in EHR
8. Diagnosed with medical condition likely to be terminal within 24 weeks as documented in EHR
9. On wait list for heart transplantation or ventricular assist device (VAD) as documented in EHR
10. NYHA Stage IV HF or end-stage COPD as documented in EHR
11. Receiving hospice care as documented in EHR
12. Active substance abuse as documented in EHR
13. Has end stage renal disease or is currently receiving dialysis

Qualitative Interview Exclusion Criteria

1. Randomized to the control arm

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Comparison of actual and anticipated recruitment rates | 30 days post discharge
  Actual rates of recruitment as compared to the anticipated recruitment rate of at least 35% of those approached for the study.
Comparison of actual and anticipated retention rates | 30 days post discharge
  Actual rates of retention as compared to the anticipated retention rate of 70% of participants until the final survey time point.
Comparison of actual and anticipated attendance rates | 30 days post discharge
  Actual rates of attendance rates as compared to the anticipated 3/4 sessions among at least 70% of participants in the music therapy arm.
Comparison of actual and anticipated completion rates | 30 days post discharge
  Actual rates of completion rates as compared to the anticipated at least 70% of 15-day and 30-day follow-up measures.
Number of participants report daily music exercise use | 30 days post discharge
  At least 60% of participants in the music therapy arm reporting use of music exercises at least once every other day.
Acceptance of music therapy intervention | 37 days post discharge
  Favorable responses to qualitative interviews

SECONDARY OUTCOMES:
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Physical function (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Anxiety (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Depression (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Fatigue (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Sleep disturbance (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Ability to participate in social roles and activities (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Pain interference (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) General Self Efficacy - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  General self-efficacy (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Emotional support (4 questions)
Change from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Instrumental Support - Short Form 4a | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Instrumental support (4 questions)
Change from baseline in Perceived Stress Scale - 4 | Pre-test at baseline, 15 days post-discharge, and 30 days post-discharge
  Perceived stress (4 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodgers-Melnick, MPH, MT-BC, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No